



# Cover Page

## 1. Official Title of the Study

An international study on the professional quality of life of youth care workers.

## 2. NCT Number

Not yet assigned

## 3. **Document Type**

Study Protocol with Statistical Analysis Plan (SAP)

## 4. Version and Document Date

Version 8 - 17/05/2024





## Study Protocol

Study Title: An international study on the professional quality of life of youth care workers.

Protocol Version and Date: version 8, 17/05/2024

Coordinating/Principal Investigator: Prof. dr. Johan Vanderfaeillie and Camille Verheyden

## 1. Coordinating Investigator Information

Coordinating Investigator: Prof. Dr. Johan Vanderfaeillie

Principal Investigator: Camille Verheyden

Co-investigators: Renate Buisman, Edith Gorlee, Stéphanie Chartier, Séverine Euillet, Victoria Baur, Debora Caudenberg, Anke Arlette Dekeyser, Elise Eerdekens, Jana Calleja, Demi De Smet, Laura Van Den Driessche, Imke Duwé, Jasmien De Bondt, Laure Jacobs, Lien Timmers, Marthe De Smedt, Elona Vaeyens, Niels Roelant, An-Sofie Nevens, Jaber Bouyrden, Soumia El Makrini and Leila Missaoui.

Study sites and co-investigators: Vrije Universiteit Brussel, Université Liège, Université Paris Nanterre, Universiteit Leiden and Veilig Thuis Hollands-Midden.

## 2. Protocol Version History

| Version No. & date | Approval Date Lead EC |
|--------------------|----------------------------------------------|
| 1 - 12/11/2021 | Preliminary advice with remarks on 8/12/2021 |
| 2 - 16/12/2021 | Single opinion positive advice on 22/12/2021 |
| 3 - 15/02/2022 | Approval amendment A on 23/02/2022 |
| 4 - 31/03/2022 | Approval amendment B on 25/05/2022 |
| 5 - 23/11/2022 | Approval amendment C on 19/04/2023 |
| 6 - 11/05/2023 | Approval amendment D on 12/05/2023 |
| 8 - 17/05/2024 | Approval amendment E on 22/05/2024 |

## 3. Introduction

Due to their daily work with traumatized minors and their families, youth care workers (such as foster care counsellors, context counsellors, residential group workers, social workers, etc.) operate on the front line of psychologically demanding work and are frequently exposed to high levels of stress (Middleton & Potter, 2015; Boyas & Wind, 2010; Conrad & Kellar–Guenther, 2006). Youth care workers therefore represent a particularly vulnerable group for developing emotional exhaustion (Rienks, 2020). An increased risk of compassion fatigue may be the cost of their efforts and caregiving responsibilities (Middleton & Potter, 2015; Prost & Middleton, 2020; Dagan et al., 2016; Verheyden et al., 2020). In addition to the impact on personal wellbeing, these high psychological demands can significantly affect the quality of care and may influence the intention to leave the youth care profession (Middleton & Potter, 2015; Chen et al., 2012; Mor Barak et al., 2006). A high degree of emotional exhaustion thus has consequences not only for the care worker but also for youth care organizations and the clients who require continuous support. This aligns with one of the most important objectives of Flemish youth care: ensuring continuity, flexibility, and quality of the care pathway without disruptions (Flemish Integrated Youth Care Decree, 2014).

In recent years, there has been increasing interest in the *Professional Quality of Life* (ProQOL) of care professionals (Stamm, 2010). This concept captures overall psychological wellbeing and Version 8.0, 17/05/2024

2/10 | Page





the positive and negative emotions associated with caregiving work. Both positive and negative factors from the personal, client-related, and work-related domains influence a care worker's ProQOL (Stamm, 2010). ProQOL consists of two components: compassion satisfaction and compassion fatigue, which may occur simultaneously (Stamm, 2010).

Compassion satisfaction refers to the pleasure experienced by care workers when they perform their work well and can help others. Compassion fatigue is an umbrella term describing the negative emotional impact of caregiving and consists of two distinct phenomena (Adams et al., 2006; Stamm, 2010): burnout and secondary traumatic stress (STS).Burnout is associated with severe emotional and physical exhaustion, emotional and cognitive dysregulation, and mental distancing. Depressive feelings and psychological or psychosomatic tension symptoms may also occur (Schaufeli et al., 2020). This psychological condition is not immediately visible to the individual and develops gradually due to chronically demanding work situations (Schaufeli & Bakker, 2007; Figley, 1995; Lizano & Mor Barak, 2012; Maslach et al., 2001; Stamm, 2010). STS may arise from work-related secondary exposure to individuals who have experienced traumatic events. The negative symptoms related to STS parallel those of primary exposure, including anxiety, sleep problems, recurrent intrusive images, and avoidance (Stamm, 2010). Multiple studies have found a strong relationship between STS and burnout. Although both constructs originate in the work environment and show some overlap in symptom perception and expression, they are considered two distinct constructs (Stamm, 2010; Rienks, 2020; Salloum et al., 2015).

Despite the exponential growth of the integrated youth care sector and the increasing number of children and families that care services must support each year (Intersectional Annual Report, 2019), to date, little to no research has examined ProQOL and turnover intention among youth care staff in integrated youth care. Existing literature on compassion fatigue among care professionals is more extensive in the United States and the United Kingdom. For example, Rienks (2020) reported that 29.6% of U.S. youth care workers experienced severe STS and 27.3% moderate—to—high STS. Another study among the same target group (Salloum et al., 2015) found that one in three respondents experienced high levels of burnout and STS, and low levels of compassion satisfaction. Conrad and Kellar–Guenther (2006) reported that U.S. child protection workers showed significantly high levels of compassion fatigue, low burnout, and moderate compassion satisfaction. Cornille and Meyers (1999) found that 37% of child protection workers experienced clinically elevated emotional distress related to STS. Hannah and Woolgar (2018), studying British foster carers, found that 25.2% reported high STS, 30.5% high burnout, and 18.3% high compassion satisfaction.

Only limited research has examined the prevalence and risk factors of compassion fatigue in Europe or Belgium specifically. Verheyden et al. (2020) conducted the first study exploring ProQOL among Flemish foster care workers during the COVID-19 lockdown, finding low levels of STS, moderate levels of burnout, and moderate levels of compassion satisfaction. No alarming levels were observed; however, the authors noted that the findings were limited to one organization under exceptional circumstances.

With the present study, we aim to contribute to the limited body of knowledge on ProQOL, its predictors, and its relationship with turnover intention. Various organizations within integrated youth care (e.g., CKGs, foster care services, CAWs) and different types of youth care workers (e.g., foster carers, context workers, residential care workers) all face similar organizational pressures while also





experiencing individual challenges specific to their professional roles. The importance of this study lies in mapping both similarities and differences across groups and creating a foundation for future prevention and intervention efforts.

By focusing on three central study themes, we aim to generate targeted comparisons between groups, identify problem areas contributing to compassion fatigue, identify strengths associated with compassion satisfaction, and examine the link with intention to leave the youth care sector.

## 4. Study Objectives

#### a. Primary Objective

The primary objective of this study is to map the levels of secondary traumatic stress (STS), burnout, and compassion satisfaction among youth care workers employed within the Flemish integrated youth care system and to compare these levels with reference groups in Wallonia, France, and the Netherlands.

#### b. Secondary Objectives

A second objective is to identify the risk and protective factors associated with the aforementioned constructs, to examine the relationship between these constructs and the intention to leave the profession, and to compare the presence of the constructs across different target groups within Flemish youth care workers.

## 5. Intervention

The study will be conducted using an online questionnaire developed in Qualtrics. Participants may complete the questionnaire at home, and completion takes approximately 15 to 20 minutes. The questionnaire is preceded by a detailed informed consent form (see Section 8.3), and participants may only proceed to the questionnaire after providing informed consent.

The online questionnaire is organized thematically according to personal, work-related, and client-related items. After these three domains have been assessed, the outcome measures *ProQOL* and *turnover intention* are presented.

The following data will be collected in the questionnaire:

- Personal domain: Age, gender, ethnicity, partner status, children (number, relationship, gender, and whether they live at home), highest obtained degree, educational background, subjective perception of financial situation (Financial Need Scale by Ponnet et al., 2013), self-care (11 items from the Professional Self-Care Scale by Dorociak et al., 2017, and 4 items from Trauma-Informed Self-Care by Salloum et al., 2015, as used in Bridger et al., 2020), personality traits (Ten-Item Personality Inventory; Gosling et al., 2003), social support (Brief Form of the Perceived Social Support Questionnaire; F-SozU K-6 by Kliem et al., 2015), and personal trauma history.
- Work environment: Work-family conflict, quantitative workload, organizational support, support from colleagues and friends/family (General Questionnaire for Psychological and Social Factors at Work; QPS-Nordic by Elo, Dallner, Gamberale et al., 2000), organization





of employment, province of employment, distance to workplace, professional role, caseload (number of cases), professional experience (years in current role, years as youth care worker, years within the organization), and employment rate.

- Client environment: Client age category, client gender, working with clients in crisis/urgent trajectories, client trauma history (number and type of main trauma(s), and how the youth care worker is typically informed about the trauma), difficulty level of the client and parents, and over-involvement with the client (Koeske, 1995).
- Outcome measures: The Professional Quality of Life Scale Version 5 (ProQOL) by Stamm (2010) and turnover intention (as used in Prost & Middleton, 2020).

## 6. Selection of Subjects

#### 10.1 Selection of Study Population

Flemish participants will be recruited by contacting the coordinators of various youth care organizations via email and telephone. The following organizations will be contacted: all Centres for Pupil Guidance (Centra voor Leerlingenbegeleiding), Confidential Centres for Child Abuse (Vertrouwenscentra Kindermishandeling), Youth Support Centres (Ondersteuningscentra Jeugdzorg), Centres for General Welfare (Centra Algemeen Welzijnswerk), Youth Advisory Centres (Jeugdadviescentra), facilities for children and adolescents with severe behavioural and emotional problems, observation and treatment centres, Centres for Childcare and Family Support (Centra voor Kinderzorg en Gezinsondersteuning), centres for integrated family support, mental health care centres, reception–, observation– and orientation centres, special youth care organizations, foster care services, community institutions, and the Flemish detention centre in Flanders and Brussels. These organizations will receive an invitation to participate in a master's thesis research project focusing on secondary traumatic stress, burnout, and compassion satisfaction among their employees. If an organization agrees to participate, the coordinators will receive an anonymous link to the questionnaire, which they can then distribute among their staff members.

In France, Wallonia, and the Netherlands, the researchers affiliated with Université Paris Nanterre, Université de Liège, Leiden University, and Veilig Thuis Hollands-Midden will contact the coordinators and directors of their respective foster care, residential, and ambulatory youth care services. The French-language questionnaire will also be distributed via Qualtrics.

#### 10.2 Inclusion Criteria

- (1) Adults
- (2) who have a care or support relationship with children or adolescents
- (3) who are followed by an organization within the integrated youth care system (Flanders), l'aide à la jeunesse (Wallonia), la protection de l'enfance (France), or youth care services in the Netherlands.

#### 10.3 Exclusion Criteria

- (1) Adults
- (2) who have a care or support relationship with children or adolescents followed by an organization





within the integrated youth care system (Flanders), l'aide à la jeunesse (Wallonia), la protection de l'enfance (France), or Dutch youth care

(3) in cases where the likelihood of trauma exposure in the child is lower: services with a preventive character, or when the child/adolescent is followed due to a disability.

## 7. Data Collection and Management

#### a. Data Collection

Qualtrics will be used to collect the data online and anonymously. After completion of the data collection phase, the data will be analyzed in SPSS. The data will be stored in a protected folder on the VUB SharePoint environment.

b. Statistical Considerations and Data Analysis

For data analysis, IBM SPSS Statistics version 27 will be used.

First, the dataset will be screened for missing data and outliers. If necessary, cases with missing data or outliers will be removed.

To examine the levels of burnout, secondary traumatic stress, and compassion satisfaction, descriptive analyses will be performed. Comparisons with the reference groups will be conducted by means of t-tests.

To determine the risk and protective factors associated with burnout, secondary traumatic stress, and compassion satisfaction, Pearson correlation analyses, t-tests, and ANOVAs will be conducted initially. In a second step, three multiple linear regression analyses will be performed:

- 1. the first with burnout as the dependent variable and all independent variables with a significant association ( $p \le .10$ ),
- 2. the second with STS as the dependent variable and the independent variables with a significant association, and
- 3. the third with compassion satisfaction as the dependent variable and the independent variables with a significant association.

The relationship between STS, burnout, and compassion satisfaction on the one hand and turnover intention on the other hand will be examined through hierarchical regression analyses.

Using t-tests and ANOVAs, the presence of the constructs will be compared across the different target groups within integrated youth care.

## 8. Ethical Considerations

a. Ethical conduct of the study

The questionnaire will be completed anonymously via Qualtrics. The data obtained will be used exclusively for the purposes of the study and will remain confidential. Each participant will remain fully anonymous in the publication of the results. The collected data will be stored in a password-protected SharePoint folder.

#### b. Ethics Committee





The study will be submitted for approval to the Medical Ethics Committee of UZ Brussel (<a href="mailto:ethiek@uzbrussel.be">ethiek@uzbrussel.be</a>).

#### c. Informed Consent

Information letters in Dutch- and French will be provided, accordingly.

#### 8.3 Subject Identification

Because an anonymous Qualtrics link is used, responses cannot be linked to an individual person. The question regarding the organization in which the respondent is employed is used solely for calculating the response rate. Once all responses have been collected and the response rate has been calculated, this information will be removed.

Although Qualtrics normally records IP addresses, this function can be disabled. This feature is disabled in the current study to guarantee the anonymity of participants.

## 9. Reporting and Dissemination

A master's thesis will be written based on the collected data by Victoria Baur, Debora Caudenberg, Anke Arlette Dekeyser, Elise Eerdekens, Jana Calleja, Demi De Smet, Laura Van Den Driessche, Imke Duwé, Jasmien De Bondt, Laure Jacobs, Lien Timmers, Marthe De Smedt, Elona Vaeyens, Niels Roelant, An-Sofie Nevens, Jaber Bouyrden, Soumia El Makrini, and Leila Missaoui, master's students in Clinical Psychology at Vrije Universiteit Brussel. Additionally, a doctoral dissertation will be written by Camille Verheyden. The French, Walloon, and Dutch researchers will publish scientific articles based on the French, Walloon, and Dutch datasets, respectively.

## 10. Conflict of interest statement

There is no conflict of interest.





## 11. References

- Adams, R. E., Boscarino, J. A. & Figley, C. R. (2006). Compassion fatigue and psychological distress among social workers: A validation study. *American Journal of Orthopsychiatry*, 76(1), 103–108. https://doi.org/10.1037/0002-9432.76.1.103
- Borntrager, C., Caringi, J. C., van den Pol, R., Crosby, L., O'Connell, K., Trautman, A. & McDonald, M. (2012). Secondary traumatic stress in school personnel. *Advances in School Mental Health Promotion*, *5*(1), 38–50. https://doi.org/10.1080/1754730x.2012.664862
- Boyas, J. & Wind, L. H. (2010). Employment-based social capital, job stress, and employee burnout:

  A public child welfare employee structural model. *Children and Youth Services Review*,

  32(3), 380-388. <a href="https://doi.org/10.1016/j.childyouth.2009.10.009">https://doi.org/10.1016/j.childyouth.2009.10.009</a>
- Bridger, K., Binder, J., & Kellezi, B. (2020). Secondary traumatic stress in foster carers: Risk factors and implications for intervention. *Journal of Child and Family Studies*, 29(2), 482-492.
- Chen, Y. Y., Park, J. & Park, A. (2012). Existence, relatedness, or growth? Examining turnover intention of public child welfare caseworkers from a human needs approach. *Children and Youth Services Review*, 34(10), 2088–2093. https://doi.org/10.1016/j.childyouth.2012.07.002
- Conrad, D. & Kellar-Guenther, Y. (2006). Compassion fatigue, burnout, and compassion satisfaction among Colorado child protection workers. *Child Abuse & Neglect*, *30*(10),1071-1080. https://doi.org/10.1016/j.chiabu.2006.03.009
- Cornille, T. A. & Meyers, T. W. (1999). Secondary traumatic stress among child protective service workers: Prevalence, severity and predictive factors. *Traumatology*, *5*(1). https://doi.org/10.1177/153476569900500105
- Dagan, S. W., Ben-Porat, A. & Itzhaky, H. (2016). Child protection workers dealing with child abuse:

The contribution of personal, social and organizational resources to secondary traumatization. *Child Abuse & Neglect*, *51*, 203–211.

https://doi.org/10.1016/j.chiabu.2015.10.008

Decreet Integrale Jeugdhulp, 2014. Retrieved from: <a href="https://www.jeugdhulp.be/over-jeugdhulp">https://www.jeugdhulp.be/over-jeugdhulp</a>
Elo, A.-L., Dallner, M., Gamberale, F., Hottinen, V., Knardahl, S., Lindström, K., Skogstad, A., &





- Ørhede, E. (2000). Validation of the Nordic Questionnaire for Psychological and Social Factors at Work—QPSNordic. In M. Vartiainen, F. Avallone, & N. Anderson (Eds.), *Innovative theories, tools, and practices in work and organizational psychology* (pp. 47–57). Hogrefe & Huber Publishers.
- Figley, C. (1995). Compassion fatigue as secondary traumatic stress disorder: An overview. In C. Figley (Ed.), Compassion fatigue: Coping with secondary traumatic stress disorder in those who treat the traumatized (pp. 1–20). Routledge.
- Gosling, S., Rentfrow, P., & Swann, W. (2003). A very brief measure of the Big-Five personality domains. *Journal of Research in Personality*, 37(6), 504-528.
- Hannah, B. & Woolgar, M. (2018). Secondary trauma and compassion fatigue in foster carers.

  \*\*Clinical Child Psychology and Psychiatry, 23(4), 629-643.\*\*

  https://doi.org/10.1177/1359104518778327
- Kliem, S., Mößle, T., Rehbein, F., Hellmann, D. F., Zenger, M., & Brähler, E. (2015). A brief form of the Perceived Social Support Questionnaire (FSozU) was developed, validated, and standardized. Journal of Clinical Epidemiology, 68, 551–562. http://dx.doi.org/10.1016/j.jclinepi.2014.11.003
- Koeske, G. F. & Kelly, T. (1995). The impact of overinvolvement on burnout and job satisfaction.

  \*American Journal of Orthopsychiatry, 65(2), 282–292. https://doi.org/10.1037/h0079622
- Lizano, E., & Mor Barak, M. (2012). Workplace demands and resources as antecedents of job burnout among public child welfare workers: A longitudinal study. *Children and Youth Services Review*, 34(9),1769–1776.
- Maslach, C., Schaufeli, W., & Leiter, M. (2001). Job burnout. *Annual Review of Psychology*, 52, 397-422.
- Middleton, J. S. & Potter, C. C. (2015). Relationship Between Vicarious Traumatization and

  Turnover Among Child Welfare Professionals. *Journal of Public Child Welfare*, 9(2), 195–216. https://doi.org/10.1080/15548732.2015.1021987
- Mor Barak, M. E., Levin, A., Nissly, J. A. & Lane, C. J. (2006). Why do they leave? Modeling child welfare workers' turnover intentions. *Children and Youth Services Review*, 28(5), 548-577.





- Prost, S. G. & Middleton, J. S. (2020). Professional quality of life and intent to leave the workforce:

  Gender disparities in child welfare. *Child Abuse & Neglect*, *110*, 104535.

  https://doi.org/10.1016/j.chiabu.2020.104535
- Rienks, S. L. (2020). An exploration of child welfare caseworkers' experience of secondary trauma and strategies for coping. *Child Abuse & Neglect*, *110*, 104355.

  https://doi.org/10.1016/j.chiabu.2020.104355
- Salloum, A., Kondrat, D. C., Johnco, C. & Olson, K. R. (2015). The role of self-care on compassion satisfaction, burnout and secondary trauma among child welfare workers. *Children and Youth Services Review*, 49, 54-61. https://doi.org/10.1016/j.childyouth.2014.12.023
- Schaufeli, W.B. & Bakker A.B. (2007). Burnout en bevlogenheid [Burnout and work engagement]. In W.B. Schaufeli & A.B. Bakker (Red.). *De psychologie van arbeid en gezondheid* (pp. 341–358). Bohn Stafleu van Loghum.
- Schaufeli, W. B., Desart, S. & De Witte, H. (2020). Burnout Assessment Tool (BAT)—Development,

  Validity, and Reliability. *International Journal of Environmental Research and Public Health*,

  17(24), 9495. <a href="https://doi.org/10.3390/ijerph17249495">https://doi.org/10.3390/ijerph17249495</a>
- Sprang, G., Craig, C., & Clark, J. (2011). Secondary traumatic stress and burnout in child welfare workers: a comparative analysis of occupational distress across professional groups. *Child welfare*, 90(6), 149–68.
- Stamm, B. H. (2010). The concise ProQOL manual. Pocatello, ID: <a href="mailto:ProQOL.org">ProQOL.org</a>; Retrieved from <a href="http://ProQOL.org/uploads/ProQOL\_Concise\_2ndEd\_12-2010.pdf">http://ProQOL.org/uploads/ProQOL\_Concise\_2ndEd\_12-2010.pdf</a>
- Verheyden, C., Van Holen, F., West, D. & Vanderfaeillie, J. (2020). Secondary traumatic stress, burnout and compassion satisfaction among Flemish foster care workers during the COVID-19 lockdown. *Developmental Child Welfare*, 2(4), 227-243. https://doi.org/10.1177/2516103220987227
- Vlaamse jeugdhulp, Intersectoraal jaarverslag, 2019. Retrieved from:

  https://www.jaarverslagjeugdhulp.be/over-jeugdhulp/over-jeugdhulp-uitgebreide-tekst